CLINICAL TRIAL: NCT02338856
Title: A Phase I Clinical Trial to Evaluate the Pharmacokinetics and Safety of MB12066 in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetic Study of MB12066 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: MB12066_003
Record Dates: First submitted 2015-01-11; First posted 2015-01-14 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Metabolic Syndrome
Keywords: Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — beta-lapachone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MB12066 200mg (Experimental)
  Interventions: Drug: MB12066 200mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB12066 200mg — 100mg bid (multiple dose, day 8)
  Arms: MB12066 200mg
Drug: Placebo — 100mg bid (multiple dose, day 8)
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of MB12066 after multiple dose and to investigate the pharmacokinetic characteristics of MB12066 after multiple dose.

ELIGIBILITY:
Inclusion Criteria:

* Subject is informed of the investigational nature of this study and voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) - approved informed consent prior to performing any of the screening procedures
* Healthy Korean male volunteers, age ranged 20 to 45 years
* A subject with body weight between 60 kg (inclusive) and 90 kg (exclusive) and body mass index (BMI) between 18.5 (inclusive) and 25 (exclusive). ☞ BMI (kg/m2) = weight (kg) / {height (m)}2
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the laboratory reference ranges for the relevant laboratory tests (unless the investigator considers the deviation to be irrelevant for the purpose of the study)

Exclusion Criteria:

* A subject with history of allergies including drug allergies (aspirin, antibiotics, etc.), or history of clinically significant allergies
* A subject with clinical evidence or history of hepatic (including carrier of hepatitis virus), renal, respiratory, endocrine, neurologic, immunologic, hematologic, oncologic, psychiatric, or cardiovascular disease
* A subject with history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
* A subject whose hemoglobin(Hb) level < 12 g/dL
* A subject with fasting plasma glucose (FPG) level < 70 mg/dL or ≥ 126 mg/dL
* A subject whose systolic blood pressure (SBP) ≤ 90 mmHg or ≥ 140 mmHg, diastolic blood pressure (DBP) ≤ 40 mmHg or ≥ 90 mmHg or pulse rate (PR) ≥ 100 /min after at least 5 min sitting
* A subject with history of drug abuse
* A subject who has taken any prescribed medication or herbal compounds within 14 days prior to the study drug administration. In addition, a subject who has taken any over-the-counter drug or vitamin supplements within 7 days prior to the study drug administration (However, investigators can judge the subject, who has taken the medications during those periods above, eligible for the trial if all other conditions are satisfied.)
* A subject who has participated in any other clinical trial either for investigational or marketed drugs within 8 weeks before the study drug administration
* A subject who has donated or had loss of ≥ 400 mL of blood within 8 weeks prior to start of administration of study drug
* A subject who consumes more than 21 units of alcohol per week or unable to stop drinking throughout the study period
* A smoker (except for whom quitted smoking prior to the drug administration for at least 3 months)
* A subject who heavily takes caffeine or caffeine-containing products, grapefruit, grapefruit juice, grapefruit-containing products
* A subject with unusual dietary habit
* A subject who was previously assigned to treatment during this study
* The investigator judges the subject not eligible for the study after reviewing clinical laboratory results or other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of reported adverse events | from day 1 to day 14-18

SECONDARY OUTCOMES:
Composite of Pharmacokinetic parameters | day 1, day 5, day 8
  day 1 : pre-dose(0h), 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24h day 5 : pre-dose(morning) day 8 : pre-dose(0h), 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 36, 48, 60h

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook National University Hospital, Daegu, Dongduck-ro, Jung-gu, South Korea